CLINICAL TRIAL: NCT05052073
Title: Interaction of Muscle Dystrophy, Glucose Metabolism and Insulin Sensitivity
Acronym: MyoMet
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Michael Boschmann, Dr. med., Charite University, Berlin, Germany
Other Study IDs: MyoMet
Record Dates: First submitted 2021-09-09; First posted 2021-09-22 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Various Forms of Skeletal Muscle Dystrophy
Keywords: muscle dystrophy; energy metabolism; calorimetry; metabolic chamber; microdialysis; exercise
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Biospecimen Retention: Samples Without DNA — * blood sample
  * adipose tissue dialysate samples (microdialysis)
  * skeletal muscle dialysate samples (microdialysis)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MD patients: * patients with different forms of muscle dystrophy, for example
  * facioscapulohumeral dystrophy
  * dysferlinopathy
  * caveolinopathy
  Interventions: Diagnostic Test: oral glucose load at rest; Diagnostic Test: oral glucose load and exercise
- Controls: - healthy age- and sex-matched controls (10 men, 10 women)
  Interventions: Diagnostic Test: oral glucose load at rest; Diagnostic Test: oral glucose load and exercise

INTERVENTIONS:
Diagnostic Test: oral glucose load at rest — oral glucose load (75 g) after an 12h overnight fast at rest accompanied by blood sampling and dialysate sampling (adipose tissue and skeletal muscle), and calorimetry (canopy) over three hours.
Diagnostic Test: oral glucose load and exercise — oral glucose load (75 g) after an 12h overnight fast followed by a defined (0.5 W / kg), moderate bicycle exercise i a metabolic chamber

SUMMARY:
The aim of this project to characterize systemic and organ-specific (subcutaneous adipose tissue and skeletal muscle) metabolic responses at rest and during standardized, moderate exercise after an oral glucose load in patients with various geneticaly heritable foms of skeletal muscle dystrophies. Metabolic responses will be monitored by indirect calorimetry (canopy and/or metabolic chamber at rest and during exercise) and microdialysis (adipose tissue and skeletal muscle at rest) before and after an oral glucose load (75 g).

ELIGIBILITY:
Inclusion Criteria:

* controls: healthy, no metabolic, endocrine, neurologic or other diseases
* patients: genetically confirmed diagnosis of muscle dystrophy

Exclusion Criteria:

* known hemorrhagic diseases / coagulopathies
* intake of oral anti-coagulant drugs (control of PTT, INR and platelet count before study entry)
* insulin-dependent Diabetes mellitus
* pregnancy and lactation period
* chronic use of non-steroidal antiphlogistics
* alcohol and drug abuse
* Claustrophobia • gleichzeitige Teilnahme an einer anderen Studie; Teilnahme an einer Studie vor weniger als zwei Monaten Unfähigkeit, die mündlichen und schriftlichen Informationen zur Studie zu verstehen und das schriftliche Einverständnis zu geben

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * out-patient clinic at Charité Universitätsmedizin Berlin, Campus Buch
  * University Campus of Charité Universitätsmedizin Berlin
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2009-09-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
muscle dialysate lactate | 15 minutes intervals after glucose over three hours
  marker for anaerobic glycolysis
muscle dialysate pyruvate | 15 minutes intervals after glucose over three hours
  marker for aerobic glycolysis

SECONDARY OUTCOMES:
muscle tissue perfusion | 15 minutes intervals after glucose over three hours
  measured by microdialysis and ethanol dial / ethanol perf ratio (no dimensions)
energy expenditure | 15 minutes intervals after glucose over three hours
  measured by indirect calorimetry either at rest (canopy device) or during exercise (metabolic chamber)

CONTACTS AND LOCATIONS:
Locations (1):
- Charite University Medicine, ECRC, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No